CLINICAL TRIAL: NCT00997360
Title: A Phase 1 Study of PKI-179 Administered Orally to Subjects With Solid Tumors
Brief Title: Study of PKI-179 Administered Orally to Subjects With Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3266A1-1002
Record Dates: First submitted 2009-10-16; First posted 2009-10-19 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: Phase 1; Maximum tolerated dose; Solid tumors
MeSH Terms: interventions — 1-(4-(4-(3-oxa-8-azabicyclo(3.2.1)octan-8-yl)-6-morpholino-1,3,5-triazin-2-yl)phenyl)-3-(pyridin-4-yl)urea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): PKI-179
  Interventions: Drug: PKI-179

INTERVENTIONS:
Drug: PKI-179

SUMMARY:
This is an open label dose escalation study to find the maximum tolerated dose (MTD) of PKI-179 in subjects with solid tumors. Part 1 of the study will be the dose estimation phase and will be open to subjects with all solid tumors. Part 2 will be the dose confirmation phase and will be open to subjects with breast, non small cell lung, ovarian, endometrial, or colorectal cancer or glioblastoma. All subjects will receive daily oral dosing of PKI-179. A continuous reassessment method (CRM) design will be used, which will take into account dose limiting toxicity (DLT) information from each dose level explored in order to determine the next dose level.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age 18 years or older.
2. Part 1/MTD Estimation Phase: Pathologic diagnosis of any solid tumor. Part 2/MTD Confirmation Phase: Pathologic diagnosis of one of the following tumor types: breast, non-small cell lung, ovarian, endometrial, or colorectal cancer or glioblastoma.
3. Availability of either formalin-fixed paraffin-embedded (FFPE) tumor tissue block or unstained slides for exploratory biomarker analysis.
4. Incurable cancer, with disease progression following at least 1 conventional, standard, or investigational therapy with no further standard treatment available in the opinion of the investigator.
5. At least 1 evaluable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
6. Eastern Cooperative Oncology Group (ECOG) 0 to 2.
7. Acceptable laboratory values, including fasting serum glucose.
8. All male and female subjects who are biologically capable of having children, must agree to use a medically acceptable method of birth control for the duration of the study (e.g., condom with a spermicide) and for 12 weeks after the last dose of investigational product. All female subjects who are biologically capable of having children must have a negative serum pregnancy test result before first dose of investigational product. Any pregnancy that occurs in the female partner of a male subject in the trial must be reported if it occurs at any time during the active treatment phase of the study or for 12 weeks after the last dose of investigational product.

Exclusion criteria:

1. Major surgery, chemotherapy, radiotherapy, investigational therapy, or other cancer therapy within 2 weeks prior to first dose of investigational product.
2. Lack of recovery from any prior surgery, chemotherapy, radiotherapy, or other cancer therapy.
3. Clinically unstable primary or metastatic central nervous system (CNS) tumors. Subjects with progression of CNS tumors are eligible as long as they have been clinically stable for at least 4 weeks before first dose of PKI-179 (no significant change in anticonvulsant doses, mental status, or clinical symptoms related to the CNS tumors).
4. Subjects with known diabetes.
5. QTc interval > 470 ms.
6. Pregnant or breastfeeding women.
7. Evidence of significant medical illness or abnormal laboratory finding that in the opinion of the investigator would substantially increase the risk associated with the subject's participation in the study or impact the assessment of safety and/or efficacy. Examples include, but are not limited to: uncontrolled seizures, serious ongoing active infection requiring treatment, significant uncontrolled cardiac disease, such as congestive heart failure, myocardial infarction within past 6 months, angina requiring treatment, or other clinically significant or uncontrolled conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by physical examinations, electrocardiograms, laboratory assessments, vital signs, adverse events and serious adverse events | 1 year

SECONDARY OUTCOMES:
Tumor assessments, blood samples to look at how the drug enters your body and what the body does with it. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer